CLINICAL TRIAL: NCT06810622
Title: NAVIGATE CKD: A Community-engaged Multi-level Intervention to Reduce Kidney Disparities Among Latinos With Kidney Disease
Brief Title: NAVIGATE Kidney: A Multi-level Intervention to Reduce Kidney Health Disparities
Acronym: NAV-Kidney
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of New Mexico (Other); Denver Health and Hospital Authority (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-2014
Record Dates: First submitted 2024-10-18; First posted 2025-02-05 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Kidney Diseases; Chronic Kidney Diseases
Keywords: Kidney; Chronic; Dialysis; Transplant
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency, Chronic; Bronchiolitis Obliterans Syndrome | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Our clinical trial is a multi-site, unblinded, patient-level randomized controlled trial that will randomize 450 adult Latinx individuals with CKD stage 4/5 (eGFR 15-29 mL/min/1.73m2). The two arms include: (1) NAVIGATE-Kidney, a CHW Arm, in which a CHW will provide support during visits every 2 weeks for 3 months (i.e., 6 visits during first 3 months) followed by monthly visits until end of study or until 3 months following KRT start or (2) a Control (standard care) Arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAVIGATE-Kidney CHW (Other): A CHW will provide support during visits every 2 weeks for 3 months (i.e., 6 visits during first 3 months) followed by monthly visits until end of study or until 3 months following KRT start.
  Interventions: Other: Navigate-Kidney CHW
- NAVIGATE-Kidney Control (Other): Participants will receive standard medical care following diagnosis. This care will include educational materials developed that describe prevention of CKD progression, KRT options, and conservative management in English or Spanish.
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Navigate-Kidney CHW — A CHW will provide support during visits every 2 weeks for 3 months (i.e., 6 visits during first 3 months) followed by monthly visits until end of study or until 3 months following KRT start. As well as receiving educational materials that describe prevention of CKD progression, KRT options, and conservative management in English or Spanish
  Arms: NAVIGATE-Kidney CHW
Other: Standard Care — Participants will receive standard medical care as well as educational materials developed that describe prevention of CKD progression, KRT options, and conservative management in English or Spanish
  Arms: NAVIGATE-Kidney Control

SUMMARY:
The overarching goal of this project is to refine and adapt previous work on the NAVIGATE-Kidney project for Latinx with CKD. The investigators hypothesize that the multilevel NAVIGATE-Kidney program intervention will reduce the rate of central venous catheter use at KRT start (primary outcome), increase the rate of optimal KRT starts (secondary outcome), increase patient activation, and reduce decisional conflict (patient-centered outcomes) for Latinx with advanced CKD. The project will have four (4) aims.

DETAILED DESCRIPTION:
The overarching goal of this project is to eliminate structural racism and reduce kidney health disparities faced by Latinx (gender-inclusive term; includes Hispanics, Latino/a/x) individuals. The team developed Navigate-Kidney, a community health worker (CHW) intervention to improve clinical and person-centered outcomes for Latinx with kidney failure receiving maintenance hemodialysis. The investigators now aim to test NAVIGATE-Kidney among individuals with advanced CKD stage 4/5. The investigators hypothesize that compared to standard care, the multilevel NAVIGATE-Kidney intervention will reduce the composite endpoint, defined as (1) time to transition to KRT and central venous catheter use or (2) death (primary outcome), increase the rate of optimal KRT starts and optimal KRT process measures (secondary clinical outcomes), increase patient activation, reduce social challenges, and reduce decisional conflict (patient-centered outcomes) for Latinx with advanced CKD stage 4/5 (eGFR 15-29 mL/min/1.73m2). The investigators will also evaluate Navigate-Kidney implementation outcomes using the PRISM (Practical Robust Implementation and Sustainable Model) science framework and conduct an economic evaluation to inform policy change.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age,
* Adults who self-identify as Latino/e/a/x and/or Hispanic,
* Adults who are not pregnant,
* Adults who are not incarcerated,
* Adults who have advanced kidney disease with an eGFR of 15-29 mL/min/1.73m2). No other measures are used to identify eligible patients.

Exclusion Criteria:

* Anyone who does not meet the criteria outlined above.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite Outcome: Time Until Kidney Replacement Therapy (KRT) Start with Central Venous Catheter (CVC) Use or Death | From Baseline until End of Study, KRT Start, or Death, whichever occurs first (up to 5 years)
  Composite outcome of time until participants in each arm either 1) begin dialysis (either as first KRT method or as a subsequent preparatory step for transplant) with a central venous catheter (CVC)), or 2) die from all-cause mortality, whichever occurs first.

SECONDARY OUTCOMES:
Rate of Central Venous Catheter (CVC) use at onset of Kidney Replacement Therapy (KRT) or Death | From Baseline until End of Study, KRT Start, or Death, whichever occurs first (up to 5 years)
  Rate of participants in each arm that either 1) "crash start" Kidney Replacement Therapy (KRT) via first starting dialysis with a Central Venous Catheter (CVC), or 2) die from all-cause mortality prior to starting any method of KRT, whichever occurs first.
Rate of Participants with Optimal Kidney Replacement Therapy (KRT) Start | From Baseline until End of Study, KRT Start, or Death, whichever occurs first (up to 5 years)
  Rate of patients with condition: "Optimal KRT start", a composite measure (defined by the CMS Kidney Care Choices (KCC) value-based payment model) that includes patients with any of the following: 1. Pre-emptive kidney transplant; 2. Home dialysis; and/or 3. In-center dialysis start with a functional arteriovenous fistula or graft.
Time to First Optimal Kidney Replacement Therapy (KRT) Process Measure Milestone | From Baseline until End of Study, KRT Start, or Death, whichever occurs first (up to 5 years)
  Optimal Kidney Replacement Therapy (KRT) start process measure milestones are defined as the following: (1) Endpoints for permanent vascular access: vascular mapping and surgical visit or referral; (2) Endpoints for kidney transplant: Initial transplant visit, undergoing work-up for waitlisting, and waitlisting; (3) Endpoints for home dialysis: Initial evaluation visit for home dialysis.
Change in Estimated Glomerular Filtration Rate eGFR | Screening until End of Study or Death, whichever occurs first (up to 5 years)
  Measure of kidney function, reported in mg/dL. Scores of less than 15 may indicate kidney failure, while scores of 90 or higher indicate normal kidney function.
Change in Decisional Conflict Scale (DCS) scores | Baseline, Month 6, Month 12, Month 24
  Decisional Conflict Scale (DCS) is a 16-item tool that evaluates patient decisional conflict in 4 domains: informed, clarity, uncertainty, and support. Possible total scores range from 0 to 100, with higher scores indicating higher decisional conflict and worse outcomes.
Change in Patient Activation (PAM-13) scores | Baseline, Month 6, Month 12, Month 24
  Patient activation is measured with the Patient Activation Measure 13 (PAM-13), ranging in scores from 0 to 100. Higher scores are associated with improved behaviors related to the patient's self-management of their health and disease, and a better outcome.
Change in Quality of Life, as measured by Patient-Reported Outcomes Measurement Information Systems' (PROMIS) Global Health Scale scores | Baseline, Month 6, Month 12, Month 24
  The PROMIS Global Health Scale Version 1.2. is a 10-item tool that evaluates self-reported measures of patients' physical health and function. Possible scores range from 1-10, with higher scores indicating better health and function, and better outcomes.
Change in Social Determinants of Health, as measured by AHC-HRSN Responses | Baseline, Month 6, Month 12, Month 24
  The Accountable Health Communities (AHC) Health-Related Social Needs (HRSN) Screening Tool is a 10-item, tool that identifies health-related social needs (HRSNs) in patients in 5 domains: Housing Instability, Food Insecurity, Transportation Problems, Interpersonal Safety, and Utility Help needs. Each item is scored using a Yes/No response format. Yes answers indicate a positive screening for a patient need.
Change in KRT knowledge as measured by the Rotterdam Renal Replacement Knowledge Test (R3K-T, 30 items) | Baseline, Month 6, Month 12, Month 24
  The Rotterdam Renal Replacement Knowledge test (R3K-T) is a 30-item tool that assesses participant knowledge of renal replacement therapy. Possible scores range from 0 to 30, with higher scores indicating more correct answers and higher participant knowledge about therapy.
Change in Medical Mistrust, as measured by the Medical Mistrust Index (MMI) | Baseline, Month 6, Month 12, Month 24
  The Medical Mistrust Index (MMI) is an 11-item measure that evaluates participants' mistrust of health care organizations. The MMI items are scored on a 4-response Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree), with higher scores indicating more mistrust of healthcare organizations

OTHER OUTCOMES:
Dissemination and implementation RE-AIM outcomes for Navigate-Kidney | Baseline up to End of Study (up to 5 Years)
  PRISM (Practical Robust Implementation and Sustainable Model) contextual factors will be used to assess dissemination and implementation outcomes. PRISM consists of 2 parts: 1) Key contextual factors that impact implementation 2) Implementation outcomes called RE-AIM (Reach-Effectiveness-Adoption-Implementation-Maintenance).
  Qualitative interviews with community health workers and participants assigned to the NAVIGATE-Kidney intervention arm will be conducted.
Economic Evaluation Outcomes | Baseline up to End of Study (up to 5 Years)
  Estimations of the cost of implementing and sustaining the intervention, and analysis to determine the economic value of NAVIGATE-kidney by calculating the incremental cost-effectiveness ratio (ICER) compared to standard care.

CONTACTS AND LOCATIONS:
Overall Officials: Lilia Cervantes, MD, Principal Investigator — University of Colorado-Anschutz SOM-Hospital Medicine
Locations (2):
- United States (2):
  - Denver Health and Hospital Authority, Denver, Colorado
  - University of New Mexico Health Science Center, Albuquerque, New Mexico

IPD SHARING:
Plan to Share IPD: Yes
Limited data sets will be shared at end of study via an NIDDK registry: NIDDK-CR, in accordance with NIDDK data sharing policies.
Time Frame: Within 12 months of Primary Completion Date, ongoing.
URL: https://repository.niddk.nih.gov/home